CLINICAL TRIAL: NCT03900676
Title: A Phase 2, Randomized, Multicenter, Double-blind, Vehicle-controlled, Dose-ranging Study to Evaluate the Efficacy and Safety of VB-1953 Topical Gel When Applied Once or Twice Daily for 12 Weeks in Subjects With Moderate to Severe Inflammatory Facial Acne Vulgaris
Brief Title: Efficacy and Safety Study of VB-1953 Topical Gel for Inflammatory Facial Acne Vulgaris
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Vyome Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VTI/CR&MA/2019/001
Record Dates: First submitted 2019-04-01; First posted 2019-04-03 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — VB-1953

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Care Provider, Investigator
Masking Description: Triple (Participant, Care Provider, Investigator)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- VB-1953 topical gel - 2% QD (Experimental): VB-1953 topical gel - 2% QD
  Interventions: Drug: VB-1953 - 2%
- VB-1953 topical gel - 2% BID (Experimental): VB-1953 topical gel - 2% BID
  Interventions: Drug: VB-1953 - 2%
- VB-1953 topical gel- 0% (Vehicle) QD (Placebo Comparator): VB-1953 topical gel- 0% (Vehicle) QD
  Interventions: Drug: VB-1953 - 0% (Vehicle)
- VB-1953 Vehicle (Placebo Comparator): VB-1953 topical gel- 0% (Vehicle) BID
  Interventions: Drug: VB-1953 - 0% (Vehicle)

INTERVENTIONS:
Drug: VB-1953 - 2% — Topical Gel
  Arms: VB-1953 topical gel - 2% BID; VB-1953 topical gel - 2% QD
Drug: VB-1953 - 0% (Vehicle) — Topical Gel
  Arms: VB-1953 Vehicle; VB-1953 topical gel- 0% (Vehicle) QD

SUMMARY:
A Phase 2, Multicenter, Randomized, Double-Blind, Vehicle Controlled, Dose-ranging Study in the Treatment of Acne Vulgaris,

DETAILED DESCRIPTION:
This will be a Phase 2, multicenter, randomized, double-blinded, dose-ranging, parallel arm comparison study in male and non-pregnant female subjects, 9 through 45 years of age (inclusive) with facial acne vulgaris. This dose-ranging study, intended to identify the dose(s), will consist of 7 study visits over 14 weeks:

ELIGIBILITY:
Inclusion Criteria:

* Males or non-pregnant females 9 to 45 years of age (inclusive) at the time of consent/assent.
* Have a clinical diagnosis of moderate to severe (Grade 3 or 4) facial acne vulgaris, as determined by the Investigator's Global Assessment (IGA).
* Have 20 to 50 inflammatory lesions (papules, pustules) on the face.
* Have 20 to 60 non-inflammatory lesions on the face.

Exclusion Criteria:

* Has more than two (2) facial nodulocystic lesions.
* Female subject is pregnant, lactating, or is planning to become pregnant during the study.
* Has active nodulocystic acne or acne conglobata, acne fulminans, or other forms of acne (e.g., acne mechanica). In the opinion of the Investigator, the subject has a skin pathology or other medical condition that is clinically significant (e.g., obesity) and will preclude participation in the study.
* Has presence of any skin condition on the face (e.g., rosacea, dermatitis, psoriasis, squamous cell carcinoma, eczema, acnetiform eruptions caused by medications, steroid acne, steroid folliculitis, or bacterial folliculitis) in the opinion of the Investigator that could interfere with the diagnosis or assessment of acne vulgaris or evaluation of the investigational product (IP) or requires the use of interfering topical or systemic therapy.
* Not willing to minimize or avoid natural and artificial sunlight exposure during treatment.

Ages: 9 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 480 (Estimated)
Dates: Start 2019-04-09 (Actual); Primary Completion 2019-11 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Inflammatory lesion counts | 12 weeks
  Absolute Change from Baseline in inflammatory lesion counts in each treatment arm at Week 12.

SECONDARY OUTCOMES:
Investigator's Global Assessment of Inflammatory Acne (IGA) score | 12 weeks
  Proportion of subjects achieving success at Week 12, with success defined as Investigator's Global Assessment of Inflammatory Acne (IGA) score of 0 (clear) or 1 (almost clear) with at least a 2-point improvement from Baseline.
Percent change in inflammatory lesion counts | 12 weeks
  Percent change from Baseline in inflammatory lesion counts in each treatment arm at Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Shilpi Jain, Study Director — Vyome Therapeutics Inc.
Locations (11):
- United States (11):
  - Vyome Therapeutics Inc., Ontario, California
  - Vyome Therapeutics Inc., Sherman Oaks, California
  - Vyome Therapeutics Inc., Brandon, Florida
  - Vyome Therapeutics Inc., Coral Gables, Florida
  - Vyome Therapeutics Inc, Miami, Florida
  - Vyome Therapeutics Inc., Winter Park, Florida
  - Vyome Therapeutics Inc., High Point, North Carolina
  - Vyome Therapeutics Inc., Hazleton, Pennsylvania
  - Vyome Therapeutics Inc., Upper Saint Clair, Pennsylvania
  - Vyome Therapeutics Inc., Mt. Pleasant, South Carolina
  - Vyome Therapeutics Inc., El Paso, Texas

IPD SHARING:
Plan to Share IPD: No
Do not plan to share IPD.